CLINICAL TRIAL: NCT01944371
Title: Short-term Disulfiram Administration to Reverse Latent HIV Infection: a Dose Escalation Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Monash University (Other); amfAR, The Foundation for AIDS Research (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Steven Deeks, Professor of Medicine, University of California, San Francisco
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-10948; DAIDS-ES ID 11864 (Other Grant/Funding Number: NIAID); K24AI069994 (NIH)
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Results first posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2018-12

CONDITIONS: HIV; Human Immunodeficiency Virus
Keywords: Latent reservoir
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Disulfiram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- disulfiram 500mg (Experimental): 500mg disulfiram by mouth per day for 3 days
  Interventions: Drug: Disulfiram
- disulfiram 1000mg (Experimental): 1000mg disulfiram by mouth per day for 3 days
  Interventions: Drug: Disulfiram
- disulfiram 2000mg (Experimental): 2000mg disulfiram per mouth per day for 3 days
  Interventions: Drug: Disulfiram

INTERVENTIONS:
Drug: Disulfiram — This study will provide open label disulfiram. Subjects will take 1 dose of disulfiram per day for 3 days.
  Other Names: Antabuse,NDC 0093-5036-01

SUMMARY:
The purpose of this study is to determine the safety, pharmacology and bioactivity of disulfiram in antiretroviral treated HIV-infected adults. The investigators primary hypothesis is that 3 days of disulfiram will result in an increase in HIV transcription in CD4+ T-cells in patients on suppressive antiretroviral therapy (ART).

DETAILED DESCRIPTION:
Combination antiretroviral therapy for HIV-1 infection can suppress viremia to below the detection limit in the vast majority of motivated individuals with access to these drugs. However, HIV-1 persists in a small pool of latently infected resting memory CD4+ T cells carrying integrated viral genomes. Although other reservoirs for HIV-1 exist, the general consensus among experts is that latent virus (HIV DNA in resting memory CD4+ T cells) is the primary barrier to HIV-1 eradication. A widely discussed approach for eliminating this viral reservoir requires reactivation of latent HIV-1. Disulfiram, an FDA-approved drug used to treat alcoholism was shown to activate HIV-1 gene expression in vitro, suggesting that activation of latently infected cells in vivo may occur. Our primary hypothesis is that the addition of disulfiram to a stable effective antiretroviral drug regimen will result in a dose dependent increase in HIV transcription in CD4+ T-cells in HIV-1 in patients on highly active antiretroviral therapy (HAART).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Age 18 or older
* HIV plasma viral load <50 copies/ml for at least 3 years with at least one measurement per year and most recent viral load within 3 months of screening.
* Receiving combination antiretroviral therapy (at least 3 agents); subjects must be on a efavirenz-based or a ritonavir-based regimen
* Two CD4+ T cell counts greater than 350 cell/µl in the six months prior to screening
* Willing to abstain from any alcohol one day before, during the three day period in which disulfiram will be administered and the two week period immediately after disulfiram administration

Exclusion Criteria:

* Current alcohol use disorder or hazardous alcohol use
* Current use of any drug formulation that contains alcohol or that might contain alcohol, including the gelatin capsule and liquid formulations of ritonavir, ritonavir/lopinavir, amprenavir and fosamprenavir.
* Current use of tipranavir or maraviroc.
* Current use of zidovudine, stavudine or didanosine (as disulfiram potentially has potent irreversible inhibitory effects on mitochondrial metabolism and hence could exacerbate the toxicity of these drugs).
* Concurrent use of rivaroxaban ( a CYP3A metabolized medication) as the cytochrome P450 inhibitory effects of disulfiram on rivaroxaban are unknown.
* Current use of warfarin
* Patients who are intending to modify antiretroviral therapy in the next 2 weeks for any reason.
* Serious illness requiring hospitalization or parental antibiotics within preceding 3 months
* A screening hemoglobin below 12.5 g/dL
* A screening TSH consistent with Hypothyroidism
* Significant renal disease or acute nephritis
* Significant myocardial disease or diagnosed coronary artery disease
* Significant respiratory disease
* History of psychosis, seizure disorder, abnormal electroencephalogram or brain damage with significant persisting neurological deficit.
* Clinically active hepatitis as evidenced by clinical jaundice or Grade 2 or higher liver function test abnormalities.
* Hepatic cirrhosis or decompensated chronic liver disease.
* Diabetes or current hypothyroidism.
* Concurrent treatment with immunomodulatory drugs, or exposure to any immunomodulatory drug in past 16 weeks.
* Recent exposure (within the preceding 8 weeks) to any vaccine.
* Pregnant or breastfeeding women. Women of childbearing potential must have a negative serum pregnancy test at screening and agree to use a double-barrier method of contraception throughout the study period.
* Significant substance use, which in the opinion of the investigator, is likely to interfere with the conduct of the study.
* Prior or current use of disulfiram, vorinostat or other experimental agent used with the intent to perturb the HIV-1 viral reservoir
* Current use of an antiretroviral regimen which does not include either efavirenz or a protease inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Deeks, MD, Principal Investigator — University of Californa, San Francisco; Julian Elliott, MD, Principal Investigator — Monash University
Locations (2):
- San Francisco General Hospital, San Francisco, California, United States
- Alfred Hospital, Melbourne, Australia

REFERENCES:
- [Derived] Elliott JH, McMahon JH, Chang CC, Lee SA, Hartogensis W, Bumpus N, Savic R, Roney J, Hoh R, Solomon A, Piatak M, Gorelick RJ, Lifson J, Bacchetti P, Deeks SG, Lewin SR. Short-term administration of disulfiram for reversal of latent HIV infection: a phase 2 dose-escalation study. Lancet HIV. 2015 Dec;2(12):e520-9. doi: 10.1016/S2352-3018(15)00226-X. Epub 2015 Nov 17. PMID 26614966

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 34 participants screened for eligibility, we recruited 30 participants at The Alfred Hospital (Melbourne, VIC, Australia) and the San Francisco General Hospital (San Francisco, CA, USA) between September 24, 2013, and March 31, 2014.
Period: Overall Study
Arm/Group | Disulfiram 500mg | Disulfiram 1000mg | Disulfiram 2000mg
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Disulfiram 500mg | Disulfiram 1000mg | Disulfiram 2000mg | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Full Range); unit: years] | 53 [34 to 63] | 54 [40 to 65] | 51 [26 to 67] | 53 [26 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 9 | 10 | 9 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 1 | 6
  White | 6 | 9 | 7 | 22
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 5 | 15
  Australia | 6 | 4 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Cell-associated HIV RNA
Description: Fold change cell-associated HIV RNA in Total CD4 T-Cells.
Time Frame: Baseline and 3 days
Measure: Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Disulfiram 500mg | Disulfiram 1000mg | Disulfiram 2000mg
Number analyzed (Participants) | 10 | 10 | 10
Fold change | 1.7 [1.3 to 2.2] | 1.9 [1.6 to 2.4] | 1.6 [1.2 to 2.1]

2. Secondary Outcome: Plasma HIV RNA
Description: Fold change in plasma HIV RNA levels from baseline through day 3
Time Frame: Baseline and 3 days
Measure: Mean (Full Range); unit: Fold change
Arm/Group | Disulfiram 500mg | Disulfiram 1000mg | Disulfiram 2000mg
Number analyzed (Participants) | 10 | 10 | 10
Fold change | 1.50 [0.36 to 3.4] | 0.90 [0.18 to 1.7] | 1.22 [0.32 to 2.83]

3. Secondary Outcome: Proviral HIV DNA
Description: Fold change in HIV DNA levels between Baseline and Day 30
Time Frame: Baseline and 30 days
Measure: Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Disulfiram 500mg | Disulfiram 1000mg | Disulfiram 2000mg
Number analyzed (Participants) | 10 | 10 | 10
Fold change | 1.07 [0.89 to 1.28] | 0.83 [0.60 to 1.15] | 0.91 [0.77 to 1.05]

4. Other Pre Specified Outcome: Disufiram Pharmacokinetics
Description: Plasma concentrations of disulfiram were measured on dosing day 1 (hours 0, 2, and 6), day 2 (hour 0), and day 3 (hours 0, 2, and 6), as well as on postdosing days 4, 8, and 31. The area under the curve (AUC) levels over 72 hours was estimated.
Time Frame: 31 days
Measure: Mean (97.5% Confidence Interval); unit: mg-hour/liter
Arm/Group | Disulfiram 500mg | Disulfiram 1000mg | Disulfiram 2000mg
Number analyzed (Participants) | 10 | 10 | 10
mg-hour/liter | 3,186 [3,140 to 3,281] | 8,386 [7,149 to 12,861] | 22,331 [18,481 to 35,102]

ADVERSE EVENTS:
Time Frame: Subjects were monitored in an outpatient clinic during the first 6 hours post-dose on days 1 and 3. At each visit, subjects were assessed for any new symptoms and vital signs. A complete blood count and complete metabolic panel were performed during screening, and then at Days 1, 2, 3, 4, 8 and 31. No evaluations were made after Day 31.
Description: The grading system for drug toxicities is located in the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification, August 2009), which can be found on the DAIDS RSC Web Site (http://rsc.tech-res.com/safetyandpharmacovigilance/.)
Arm/Group | Disulfiram 500mg | Disulfiram 1000mg | Disulfiram 2000mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 1/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Disulfiram 500mg (N=10) | Disulfiram 1000mg (N=10) | Disulfiram 2000mg (N=10)
Increased aspartate aminotransferase (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No